CLINICAL TRIAL: NCT06996561
Title: Exploring the Impact of Genetic Variations on The Clinical Efficacy of Nalbuphine in Postoperative Pain Management
Acronym: Nal
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Asma Abdus Salam (Other)
Responsible Party: Sponsor-Investigator, Dr. Asma Abdus Salam, Assistant Professor, Ziauddin University
Organization: Ziauddin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Nal-Gene123
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cholecystectomy; Hernia, Abdominal; Appendectomy; Open Colorectal Surgery; Laparatomy; Postoperative Pain; Hysterectomy; Cystectomy
Keywords: genetic variations; nalbuphine; opioids; polymorphism
MeSH Terms: conditions — Hernia, Abdominal; Pain, Postoperative | interventions — Nalbuphine; High-Throughput Nucleotide Sequencing; Exome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- nalbuphine (Experimental): Given as intravenously, 0.1-0.2 mg / kg at induction and intermittently
  Interventions: Drug: Nalbuphine Injection; Genetic: Next Generation Sequencing; Genetic: whole exome sequencing

INTERVENTIONS:
Drug: Nalbuphine Injection — Anaesthesia induction will be done with propofol (2 mg/kg) nalbuphine (0.1mg/kg) and atracurium (0.6mg/kg) intravenously. Maintenance of anaesthesia will be achieved with oxygen (O2), nitrous oxide (N2O) in 1:2 ratio and isoflurane (0.8-1%). Intermittent top up of the study drug 1-2 ml boluses will be administered if either the patient's HR or BP increased to 20 % above baseline and when other causes of tachycardia and hypertension are excluded. Timing of analgesia will be recorded. Pain will be assessed for 24 hours postoperatively using verbal rating scale (VRS) with 0 = no pain and 10 = worst pain. Sedation will be assessed as 0=no sedation, 1= mild sedation, (eye-opening on verbal commands), 2= moderate sedation (eye-opening on painful stimulus), 3= deep sedation (not waking up on pain). All patients will be prescribed paracetamol one gram IV six hourly and nalbuphine 1-2 mg IV infusion in the first 24 hours post operatively.
Genetic: Next Generation Sequencing — 5ml of blood samples by venipuncture will be obtained from the first 70 patients half an hour before extubation at the time of muscle closure. These blood samples will be processed for DNA analysis. Only the 15 samples where pain persisted despite nalbuphine administration, with a pain score remaining above 4, continuous use of rescue analgesia, or any documented opioid side effects (such as nausea, vomiting, or sedation), or the need for additional analgesia within 24 hours, will be sent for NGS analysis. These samples will undergo whole exome sequencing via NGS, based on patient parameters and pain scores, after being categorized as responders or non-responders to nalbuphine
  Other Names: NGS; whole exome sequencing; sanger's technique
Genetic: whole exome sequencing — Only the 15 samples will be sent for NGS based on patient parameters and pain scores after being categorized as responders or non-responders to nalbuphine
  Other Names: NGS; next generation sequencing

SUMMARY:
The goal of this study is to identify the genes as well as their association with Nalbuphine. This will help the investigator to identify opioid vulnerability in Pakistani population in the postoperative patients and will contribute to overcoming the opioid crisis, resulting in better and safer outcomes.

Research question is:

Is there any association between the underlying genetic variations and the analgesic efficacy of Nalbuphine in postoperative patients? The Research Objectives are

1. To identify the underlying genes in postoperative patients having pain.
2. To find an association between identified genes and nalbuphine clinical efficacy.

Procedure: After the written informed consent adult men and women will be enrolled in the study. On the day of surgery in the preoperative area, a 5 ml blood sample will be drawn before surgery and will be sent to laboratory for analysis. After routine hemodynamic monitoring in the operative room, general anesthesia will be given including nalbuphine. Standard routine anesthesia monitoring will be done and maintained while monitoring heart rate, ECG, NIBP oxygen saturation, ETCO2 and temperature. Incremental analgesia will be provided whenever needed. After extubation and shifting to recovery room the 2nd sample of blood will be taken and will be sent for analysis. Pain score, nausea vomiting, sedation, requirement of analgesia will be assessed till 24 hours postoperatively.

DETAILED DESCRIPTION:
The available data suggests that nalbuphine, tramadol, and morphine exhibit comparable efficacy in treating moderate to severe postoperative pain. However, significant individual variations exist in the analgesic response, which can be attributed to genetic differences. These are the variations that are influenced by a combination of demographic, clinical, and environmental factors with a significant contribution from genetic factors that regulate receptor function and signal transduction. Due to the limited availability of morphine, nalbuphine is an extensively used alternative for managing intraoperative and postoperative pain in many LMICs, particularly in Pakistan. While nalbuphine is clinically effective, there is a gap in understanding the molecular factors that contribute to its efficacy in this genetically distinct population. This highlights the need to investigate the genetic variability and to establish the analgesic efficacy of nalbuphine within Pakistani population. There is no molecular data from the region where the investigator belongs, which highlights the importance of genetic testing to tailor opioid therapy to individual needs, optimizing pain management while minimizing risks such as overdose or inadequate pain relief. By implementing genetics into clinical practice, the investigator can offer more personalized, effective, and safer opioid use, addressing the challenges associated with opioid therapy in diverse patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. All adult men or women
2. Age 18 to 70 years
3. ASA criteria 1,2 and 3
4. Abdomino-pelvic surgeries (open hernia repair, appendicectomy, open cholecystectomy, laparotomy, hysterectomy, cystectomy) lasting 2-4 hours

Exclusion Criteria:

1. Surgical procedure duration lasting more than 4 hours
2. Patients taking anti fungal fluconazole, anticoagulant (Warfarin or Clopidogrel) SNRI (Amitryptalline), Rifampicin or Buprenorphine,
3. History of hypersensitivity or allergy to opioids,
4. Pregnant or breastfeeding mothers,
5. History of narcotic dependency, addiction, and withdrawal
6. Patients experiencing any adverse side effects or complications during surgical procedure requiring intensive care admission
7. Refusing to participate in the study
8. Surgical procedures utilizing other modes of intraoperative analgesia e.g epidural analgesia or nerve blocks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
pain score | 24 hours postoperatively
  Zero is equivalent to no pain and 10 indicates the worst possible pain

SECONDARY OUTCOMES:
sedation score | 24 hours
  Sedation will be assessed as 0=no sedation, 1= mild sedation, (eye-opening on verbal commands), 2= moderate sedation (eye-opening on painful stimulus), 3= deep sedation (not waking up on pain).
nausea vomiting score | 24 hours postoperatively
  o as no nausea and vomiting and 3 as continous vomiting despite giving antiemetic
rescue analgesia | 24 hours postoperatively
  How much nalbuphine ( opioid) in mg was needed in 24 hours. will signify those not responding to conventional analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Talat Mirza, FCPS PhD, Study Director — Ziauddin University
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: A data sharing agreement must be signed. Consent and permission should be taken from the PI and officials of Ziauddin for further publication
URL: https://zu.edu.pk/office-of-research-innovation-and-commercialization-oric/

REFERENCES:
- [Result] Agarwal D, Udoji MA, Trescot A. Genetic Testing for Opioid Pain Management: A Primer. Pain Ther. 2017 Jun;6(1):93-105. doi: 10.1007/s40122-017-0069-2. Epub 2017 Apr 13. PMID 28409480